CLINICAL TRIAL: NCT01694589
Title: A Pilot Study of a Hedgehog Pathway Inhibitor (LDE-225) in Surgically Resectable Pancreas Cancer
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Rutgers Cancer Institute of New Jersey (Other); National Cancer Institute (NCI) (NIH); Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 071108; 0220120066 (Other: IRB Number); P30CA072720 (NIH)
Record Dates: First submitted 2012-09-24; First posted 2012-09-27 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-12

CONDITIONS: Resectable Pancreatic Cancer
Keywords: pancreatic cancer; resectable pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — sonidegib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LDE-225 (Experimental): LDE-225: dose - 800 mg, taken by mouth once daily for 2 weeks.
  Interventions: Drug: LDE-225

INTERVENTIONS:
Drug: LDE-225 — LDE-225 capsules will be administered as a fixed dose of 800 mg daily for two weeks.
  Other Names: NVP-LDE225; Erismodegib

SUMMARY:
We hypothesize that administration of LDE-225 in humans with pancreatic cancer will result in inhibition of paracrine HH signaling in the pancreatic tumor stroma while having no effect on autocrine signaling in the tumor cell compartment. Furthermore we hypothesize that treatment with LDE-225 will result in changes in the tumor stroma (decreased desmoplasia, increased vascularity) that will result in improved tumor blood flow.

The purpose of this study is to determine if, where and how LDE-225 works in pancreatic cancer. A cancer cell's growth can depend on the cells and tissue around it. The cells and tissue make chemical signals to influence the cancer's growth. This research study is evaluating LDE-225 designed to interfere with one of the growth signals causing pancreatic cancer growth.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy probable, resectable pancreatic cancer. Patients will be expected to undergo surgery a minimum of 14 days following signing consent.
* Patients must give informed consent.
* Patients must be over 18 and have an ECOG performance status ≤2 and life expectancy > 3 months.
* Patients must have normal organ and marrow function as defined below:

  * ANC ≥1,500 /µL
  * Platelets ≥100,000 /µL
  * Hemoglobin>10gm/dl
  * creatinine <1.5 X ULN
  * Plasma creatine phosphokinase (CK) < 1.5 x ULN
  * PT/PTT WNL
  * Patients may have abnormal bilirubin, which is concluded by the surgeon to be related to biliary ductal obstruction, may be included if bilirubin < 3 X ULN.
  * Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) < 2.5 x upper limit of normal (ULN).

Exclusion Criteria

* Poor surgical risk due to comorbidities or poor performance status
* Patients who have received prior treatment with a smoothened antagonist, (GDC-0449 (Genentech), IPI-926 (Infinity).
* Patients who have received chemotherapy within a period of time that is < the cycle length used for that treatment (e.g. <6 weeks for nitrosoureas, mitomycin-C) prior to starting study drug or who have not recovered from the side effects of such therapy
* Patients who have received wide field radiotherapy (including therapeutic radioisotopes such as strontium 89) ≤ 4 weeks or limited field radiation for palliation ≤ 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy.
* Patients who have received biologic therapy (e.g. antibodies) ≤ 4 weeks prior to starting study drug or who have not recovered from the side effects of such therapy
* Patients who have been treated with a targeted agent ≤ 5 t1/2 or ≤ 4 weeks (whichever is shorter) prior to starting study drug or who have not recovered from the side effects of such therapy
* Patients who have received any other investigational agents ≤ 5 t1/2 or ≤ 4 weeks (whichever is shorter) prior to starting study drug or who have not recovered from the side effects of such therapy
* Poor oral intake and/or inability to take capsules
* Impairment of gastrointestinal function or gastrointestinal disease such as Chron's Disease or Ulcerative Cholitis, short-gut syndrome, celiac sprue disease that may significantly alter the absorption of LDE225
* Urgent/emergent need for surgery (< 7 days)
* Documented cirrhotic liver disease, ongoing alcohol abuse, or known active or acute hepatitis
* Impaired cardiac function or clinically significant heart disease, including any one of the following:

  * Angina pectoris within 3 months
  * Acute myocardial infarction within 3 months
  * QTcF > 450 msec for males and > 470 msec for females on the screening ECG
  * A past medical history of clinically significant ECG abnormalities or a family history of prolonged QT-interval syndrome
  * Other clinically significant heart disease (e.g. congestive heart failure, uncontrolled hypertension, history of labile hypertension, or history of poor compliance with an antihypertensive regimen)
* Patients who have had a venous thromboembolic event (e.g., pulmonary embolism or deep vein thrombosis) requiring anticoagulation
* Presence of active infection or systemic use of antibiotics within 72 hours of enrollment.
* Significant co-morbid condition or disease which in the judgment of the Investigator would place the patient at undue risk or interfere with the study. Examples include, but are not limited to sepsis, recent significant cardiac or pulmonary disease, or other conditions.
* Known human immunodeficiency virus (HIV) positivity
* Known hypersensitivity to LDE-225, or any of the excipients in LDE-225
* Pregnant or lactating women.
* Patients who are receiving treatment with medications known to be moderate and strong inhibitors or inducers of CYP3A4/5 or drugs metabolized by CYP2B6 or CYP2C9 that have narrow therapeutic index, and that cannot be discontinued before starting treatment with LDE225. Medications that are strong CYP3A4/5 inhibitors should be discontinued at least 7 days and strong CYP3A/5 inducers for at least 2 weeks prior to starting treatment with LDE225.
* Patients who have neuromuscular disorders (e.g. inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis and spinal muscular atrophy) or are on concomitant treatment with drugs that are recognized to cause rhabdomyolysis, such as HMG CoA inhibitors (statins), clofibrate and gemfibrozil, and that cannot be discontinued at least 2 weeks prior to starting LDE225 treatment. If it is essential that the patient stays on a statin to control hyperlipidemia, only pravastatin may be used with extra caution.

  b) Patients who are planning on embarking on a new strenuous exercise regimen after initiation of study treatment. NB: Muscular activities, such as strenuous exercise, that can result in significant increases in plasma CK levels should be avoided whilst on LDE225 treatment.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 4 months after stopping study treatment.
* Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.
* Sexually active males must use a condom during intercourse while taking the drug and for 6 months after stopping treatment and should not father a child in this period.
* Patients unwilling or unable to comply with the protocol.

Step Two Adequate Fine Needle Biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-11; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Changes in mean Gli-1 levels before and after drug | 2 years
  Means and variances of the (transformed) data for samples from stroma and tumor are calculated. Data is collected from patients in pairs (with the first observation from the biopsy prior to drug and the second after surgery, and after the drug), and it is expected these two observations will be correlated. Detectable differences for a range of four correlations will be computed.

SECONDARY OUTCOMES:
Complications from surgery by time of hospital discharge up to 30 days post-operatively | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Darren Carpizo, MD, PhD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey, United States